CLINICAL TRIAL: NCT05839990
Title: Biomechanical and Elastic Properties of the Ascending Wall of the Human Aorta in Aneurysm
Brief Title: Biomechanical Properties of the Human Ascending Aortic Wall in Aneurysm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Tomsk NRMC aorta
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Ascending Aortic Aneurysm
MeSH Terms: conditions — Aneurysm, Ascending Aorta | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Active Comparator): Patients with ascending aortic aneurysm and dlatation who undergo surgical tretment
  Interventions: Procedure: Surgery
- Non-surgery (No Intervention): Patients with ascending aortic dlatation who undergo surveillance

INTERVENTIONS:
Procedure: Surgery — Replacement of the ascending aorta in case of anerysm and dilatation
  Other Names: Surgical treatment
  Arms: Surgery

SUMMARY:
The aim of the study is to analyze the efficacy of the surgical tretment in patients with ascending aortic aneurysm and dilatation. And to assess rate of negative clinical scenarios in non-oparated patients with ascending aortic dilatation

DETAILED DESCRIPTION:
Description of the procedures:

All surgical procedures will be performed via median sternotomy. During the aortic arch anastomosis, continuous, unilateral SACP using innominate artery will be employed. Unilateral SACP may be converted to bilateral ACP at the surgeon's discretion if adequate cerebral flows are not achieved or if there are concerns with cerebral oximetry measurements.

Once on CPB, the patient will be cooled to a nasopharyngeal (NP) temperature of 28-30 °C. Rectal temperature with be monitored as an additional temperature sites. Unilateral SACP will only be initiated once the target temperature has been reached. SACP via the innominate artery will be commenced with target flows of 8-10 ml/kg/min and perfusion pressure of 60-80 mmHg. Perfusion adequacy will be evaluated using measurement of blood pressure in both radial arteries and cerebral oximetry using near-infrared spectroscopy (NIRS).

After completion of the aortic hemiarch replacement, CPB will be resumed and the patient re-warmed to 36 °C prior to coming off CPB, with a = 1 °C temperature difference between temperature monitoring sites (NP and rectal).

Intraoperative information will be collected from the anesthetic record, surgical notes and perfusion records. Intraoperative data collection will include total operative time, CPB time, cross-clamp time, hypothermic cardiac arrest time, uSACP time, lowest nasopharyngeal and rectal temperature, arterial pressure in both radial arteries, perfusion rate and perfusion pressure during both of CPB and unilateral SACP, lowest hemoglobin concentration (g/L) and hematocrit (%), acid-base indices, intraoperative red blood cell transfusion (units), highest dose/agent used for intraoperative inotrope or vasopressor support. Also during the surgery will be performed NIRS and BIS-monitoring.

Postoperative data will include valuation of following indicators: mortality (hospital mortality and death from any cause); neurological injury (TIA, stroke, delirium), MRI and CT-scan only in event of postoperative stroke; acute kidney injury (creatinine level prior and 1, 2, 4 postoperative day (POD), urine output-up to 24-48 h, renal replacement therapy (dialysis); time of mechanical ventilation; re-exploration for bleeding, tamponade or other reasons; postoperative transfusion (packed red blood cells, platelets, fresh frozen platelets, cryoprecipitate); postoperative myocardial infarction (electrocardiogram and troponins); inotropic support during 24-48 h (agent and dose (VIS)); length of stay (intensive care unit and total hospital days).

In non-operted grop of patients annually echo cardiography, CT scans will be performed.

Aortic imaging All measurements will be taken using electrocardiography-gated computed tomographic angiography. Analysis was performed using 64-slice scanner Discovery NM-CT 570c (GE Healthcare, Milwaukee, WI, USA) with spatial resolution of the angiographic phase ranging from 0.6 to 1.25 mm. Adopted computed tomographic protocol included unenhanced, arterial, and delayed data acquisition. The arterial phase will be acquired after intravenous injection of 80-100 mL of nonionic iodinated contrast at 5 mL/s, followed by a 50-mL bolus of saline solution. Delayed-phase scans will be obtained 120-180 seconds after contrast injection. All measurements will be taken in multiplanar reconstruction, always in the plane perpendicular to the manually corrected local aortic centre line. Ascending aortic diameter will be measured at the level of the pulmonary artery bifurcation. The maximum aortic diameter (mm) will be measured from the outer contours of the aortic wall. Normalized aortic diameter (cm/m2) will be calculated by dividing the maximum aortic diameter (cm) by the body surface area (m2). The body surface area will be calculated based on the Mosteller formula: body surface area (m2) = √([Height (cm) x Weight (kg)]/3600). Analysis and assessment of the images will be based on the consensus between two experienced investigators.

Follow-up information will be collected using direct or phone contact with patients, relatives, or physicians.

ELIGIBILITY:
Inclusion Criteria:

* Ascending aortic aneurysm (50 mm and more)
* Ascending aortic dilatation (45-49 mm)

Exclusion Criteria:

* Aortic dissection
* Patients with known/documented coagulopathy
* Oncological disease (high degrees)
* Severe chronic heart failure
* Refusal of surgical treatment
* Patients in renal failure or currently being treated with renal replacement therapy (RRT) or estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2
* Severe carotid disease, defined as: any patient with previously documented carotid stenosis of > 70%, without neurological deficits; or carotid stenosis > 50% with neurological deficits; or previous carotid endarterectomy or stenting
* Pre-existing severe neurological impairment or inability to accurately assess neurocognitive function as determined by the operating surgeon

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
mortality | up to 5 years
  assess early and late death cases in aneurysm and dilatation groups in operated and nonoperarted patients
aortic growth | up to 5 years
  assess of the aortic growth in mm during foloow up in nonoperated patients

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry S Panfilov, PhD, MD, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medic
Locations (1):
- Tomsk NRMC, Tomsk, Russia